CLINICAL TRIAL: NCT04209361
Title: Assessment of Knowledge, Attitude and Practice (KAP) of Dentists at Military Hospitals Regarding Child Abuse and Neglect: A Cross-sectional Study
Brief Title: Knowledge, Attitude and Practice of Dentists at Military Hospitals Regarding Child Abuse and Neglect.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, begad hamdy ahmed own, Principal Investigator, Cairo University
Other Study IDs: Dentists and child abuse
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Child Abuse; Child Maltreatment
Keywords: Child abuse; Dentists
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Data will be obtained through a printed questionnaire for assessment of knowledge, attitude and practice of dentists at military hospitals regarding child abuse and neglect. The collected data will be saved and tabulated on a computer and finally will be statistically analyzed.

SUMMARY:
Gaining information about the knowledge, attitude and practice of dentists regarding child abuse and neglect will help identifying the points of weakness, improving their knowledge and assessing the need for additional training in relation to child protection. Thus, highlighting the importance of reporting cases of suspected child abuse which in turn may improve the status of abused children and save them from horrible situations.

DETAILED DESCRIPTION:
Children are considered to be more vulnerable than other society members because of their young age and lack of adequate skills. The annual report of United Nations Children's Fund (UNICEF) stated that a number of children have lost their lives as a result of maltreatment and violence.

Child abuse is a meaningful problem that exists among different cultural and socio-economic groups. Child abuse includes several conditions that threaten and harms lives of children. It is considered to be one of the largest causes of pediatric mortality.

The World Health Organization (WHO) defines CAN as 'Every kind of physical, sexual, emotional abuse, neglect or negligent treatment, commercial or other exploitation resulting in actual or potential harm to the child's health, survival, development, or dignity in the context of a relationship of responsibility, trust or power'.

The American Academy of Pediatric Dentistry (AAPD) defined dental neglect, as 'willful failure of a parent or guardian to seek and follow through with whatever treatment is necessary to ensure a level of oral health essential for adequate chewing function and freedom from pain and infection'.

The Child Abuse Committee of the Council on Clinical Affairs developed that definition and it was approved in 1983.

In West and Central Africa, children are susceptible to various hazards since birth including human trafficking, child labor, child marriage, conflict and other emergencies.

Frequently, abusive injuries comprise the face and oral cavity thus, dental providers may be the first to encounter these injuries. Many surveys revealed that 50 -77% of child abuse cases involving head and neck regions, consequently placing oral health care workers in an important position to detect, diagnose, document, and report to convenient authorities.

As approximately 50% of injuries due to child abuse occur in head and neck region, medical and dental professionals are in a good position for early detection and diagnosis of physical child abuse. Almost 15% of child abuse related injuries are confined to the head region Therefore, dentists have a significant role in improving the status of abused children and saving them from their dire situation.

Research has shown that guardians or parents who abuse their children regularly change their child's physicians, but very rarely change their dentists, thus dentists are considered to be in the most ideal position for detection of physical abuse in children. The American Dental Association reported the first documented evidence of dentists failing to report child maltreatment in 1967, declaring that none of 416 reported cases of child abuse was reported by a dentist in New York State.

In Egypt, few studies have discussed the problem of child abuse. Cases in most of these studies were collected from emergency, clinical departments, social welfare, criminal records or autopsies. Child abuse among Egyptian primary-school children was studied in 1994 and 1999. No data were collected regarding the prevalence of abuse among older preparatory-school and secondary school children.

Also few data are available about the knowledge, attitudes and practices of primary health care professionals toward prevention and treatment of childhood unintentional injuries.

ELIGIBILITY:
Inclusion Criteria:

* Army officer dentists at military hospitals.
* Civilian dentists at military hospitals.

Exclusion Criteria:

* Under graduate students and interns.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dentists working in military hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
knowledge, attitude and practice of dentists at military hospitals regarding child abuse and neglect. | 1 year
  Obtaining information about the knowledge, attitude and practice of dentists regarding child abuse and neglect by a printed questionnaire with binary and multiple choice questions as measuring units.

REFERENCES:
- [Background] Afifi ZE, El-Lawindi MI, Ahmed SA, Basily WW. Adolescent abuse in a community sample in Beni Suef, Egypt: prevalence and risk factors. East Mediterr Health J. 2003 Sep-Nov;9(5-6):1003-18. PMID 16450531
- [Background] Badam RK, Sownetha T, Babu DBG, Waghray S, Reddy L, Garlapati K, Chavva S. Virtopsy: Touch-free autopsy. J Forensic Dent Sci. 2017 Jan-Apr;9(1):42. doi: 10.4103/jfo.jfds_7_16. PMID 28584475
- [Background] Bunney PE, Zink AN, Holm AA, Billington CJ, Kotz CM. Orexin activation counteracts decreases in nonexercise activity thermogenesis (NEAT) caused by high-fat diet. Physiol Behav. 2017 Jul 1;176:139-148. doi: 10.1016/j.physbeh.2017.03.040. Epub 2017 Mar 28. PMID 28363838
- [Background] Definition of Dental Neglect. Pediatr Dent. 2017 Sep 15;39(6):13. No abstract available. PMID 29179302
- [Background] Fisher-Owens SA, Lukefahr JL, Tate AR; AMERICAN ACADEMY OF PEDIATRICS, SECTION ON ORAL HEALTH; COMMITTEE ON CHILD ABUSE AND NEGLECT; AMERICAN ACADEMY OF PEDIATRIC DENTISTRY, COUNCIL ON CLINICAL AFFAIRS, COUNCIL ON SCIENTIFIC AFFAIRS; AD HOC WORK GROUP ON CHILD ABUSE AND NEGLECT. Oral and Dental Aspects of Child Abuse and Neglect. Pediatrics. 2017 Aug;140(2):e20171487. doi: 10.1542/peds.2017-1487. PMID 28771417
- [Background] Hazar Bodrumlu E, Avsar A, Arslan S. Assessment of knowledge and attitudes of dental students in regard to child abuse in Turkey. Eur J Dent Educ. 2018 Feb;22(1):40-46. doi: 10.1111/eje.12242. Epub 2016 Oct 13. PMID 27735105
- [Background] Jahanimoghadam F, Kalantari M, Horri A, Ahmadipour H, Pourmorteza E. A Survey of Knowledge, Attitude and Practice of Iranian Dentists and Pedodontists in Relation to Child Abuse. J Dent (Shiraz). 2017 Dec;18(4):282-288. PMID 29201972
- [Background] Kaur H, Chaudhary S, Choudhary N, Manuja N, Chaitra TR, Amit SA. Child abuse: Cross-sectional survey of general dentists. J Oral Biol Craniofac Res. 2016 May-Aug;6(2):118-23. doi: 10.1016/j.jobcr.2015.08.002. Epub 2015 Sep 4. PMID 27195209
- [Background] Deshpande A, Macwan C, Poonacha KS, Bargale S, Dhillon S, Porwal P. Knowledge and attitude in regards to physical child abuse amongst medical and dental residents of central Gujarat: a cross-sectional survey. J Indian Soc Pedod Prev Dent. 2015 Jul-Sep;33(3):177-82. doi: 10.4103/0970-4388.160344. PMID 26156270